CLINICAL TRIAL: NCT00786838
Title: A Single-Blind, Multicenter, Placebo-Controlled, Sequential Design Study Evaluating the Potential Effects of a Single-Dose Administration of Trabectedin on the QT Intervals of the Electrocardiogram
Brief Title: A Study to Assess the Potential Effects of a Single-Dose Administration of Trabectedin on the QT Intervals of the Electrocardiogram
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Collaborators: PharmaMar (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: CR014917; ET743OVC1001 (Other: Johnson & Johnson Pharmaceutical Research and Development, L.L.C)
Record Dates: First submitted 2008-11-04; First posted 2008-11-06 (Estimated); Results first posted 2014-01-23 (Estimated); Last update posted 2014-04-11 (Estimated); Status verified 2014-03

CONDITIONS: Solid Tumor
Keywords: Solid tumor; Advanced solid tumor; Malignant tumors; Sarcoma; Breast tumor; Ovarian tumor; QT interval; Trabectedin; Yondelis; Ecteinascidin 743; ET743
MeSH Terms: conditions — Neoplasms; Sarcoma; Breast Neoplasms; Ovarian Neoplasms | interventions — Trabectedin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- Trabectedin (Experimental): 3-hour placebo intravenous infusion on Day 1 and trabectedin 1.3 mg/m2 3-hour intravenous infusion on Day 2 (single-blind). Patients may continue treatment with trabectedin until clinical benefit or drug is commercially available (open-label).
  Interventions: Drug: Trabectedin; Drug: Placebo

INTERVENTIONS:
Drug: Trabectedin — Trabectedin will be administered as 1.3 mg/m2 3-hour intravenous infusion on Day 2.
Drug: Placebo — Participants will receive 3-hour placebo intravenous infusion on Day 1.

SUMMARY:
The purpose of this study is to assess the potential effects of trabectedin on the QT/QTc interval duration measured by electrocardiograms (ECGs) in participants with advanced solid tumor malignancies when administered at a therapeutic dose.

DETAILED DESCRIPTION:
This is a single-blind (where the participant does not know the treatment he receives), multicenter (study conducted at multiple sites), placebo-controlled (an inactive substance that is compared with the study medication to test whether the study medication has a real effect in clinical study), sequential design (it is a design in a single group of Participants where one or more study medication is administered in a sequence) study to evaluate the potential effects of a single-dose administration of trabectedin on the QT intervals of the electrocardiogram (ECG). Initially, the study will consist of 2 phases: a screening phase (within 21 days before administration of the study medication), and a single-blind treatment phase (for 2 days). Participants who complete the single-blind treatment phase will be opted to take trabectedin in an open-label extension (for a minimum of 6 cycles), as long as they derive a clinical benefit (ie, until there is clear evidence of disease progression or unacceptable toxicity, as judged by the investigator). Participants will be assessed for ECG on predose before the single-blind treatment phase. During the single-blind treatment phase, a placebo control will be given on Day 1, and trabectedin (1.3 mg per square meter) will be administered on Day 2. Participants will be monitored until completion of the 24 hour pharmacokinetic blood sample collection. During the open-label extension (21 days after completion of the single-blind treatment phase), all Participants will receive trabectedin intravenously on Day 1 of each 17- to 49 day treatment cycle. The dose and schedule of trabectedin will be modified according to the type of malignancy being treated (ie, sarcoma, ovarian, or breast cancer). Safety evaluations will include assessment of adverse events, vital signs, physical examination, and clinical laboratory tests which will be performed throughout the study. The study duration for the open-label extension will vary by participant.

ELIGIBILITY:
Inclusion Criteria:

* Participants with locally advanced or metastatic solid tumors who have received three or less prior lines of systemic chemotherapy
* Participants must have relapsed or had progressive disease following standard of care treatment with chemotherapy prior to enrollment, or intolerant to prior standard of care treatment with chemotherapy
* Normal cardiac conduction and function as documented on a 12-lead electrocardiogram
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 to 1
* Adequate organ function as evidenced by laboratory tests
* Able to receive dexamethasone or its equivalent
* Agrees to protocol-defined use of effective contraception

Exclusion Criteria:

* Participants treated with more than three prior chemotherapy regimens (including adjuvant therapy)
* Previous exposure to trabectedin
* Central nervous system (CNS) metastasis
* Known hypersensitivity to any of the components of the trabectedin intravenous formulation or dexamethasone
* Heart rhythm disturbances, unusual T wave and U wave (if present) morphology, blood pressure outside of normal range, a history of cardiac failure, myocardial infarction, or cardiomyopathy, or a history of additional risk factors for torsade de pointes (eg, heart failure, electrolyte abnormalities, family history of Long QT Syndrome)
* Participants who at screening are on medication that is known to prolong the QT interval or who is on CYP3A4 inhibitors or inducers

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2008-10; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.
Locations (17):
- United States (4):
  - Miami, Florida
  - Charlotte, North Carolina
  - Philadelphia, Pennsylvania
  - Tacoma, Washington
- Belgium (3):
  - Brussels
  - Edegem
  - Wilrijk
- France (4):
  - Lyon
  - Marseille
  - Montpellier
  - Villejuif
- India (2):
  - Bengaluru
  - Pune
- Russia (2):
  - Moscow
  - Saint Petersburg
- Seoul, South Korea
- PAU de Sanchinarro, Spain

REFERENCES:
- [Derived] Thertulien R, Manikhas GM, Dirix LY, Vermorken JB, Park K, Jain MM, Jiao JJ, Natarajan J, Parekh T, Zannikos P, Staddon AP. Effect of trabectedin on the QT interval in patients with advanced solid tumor malignancies. Cancer Chemother Pharmacol. 2012 Feb;69(2):341-50. doi: 10.1007/s00280-011-1697-6. Epub 2011 Jul 8. PMID 21739119
- See also: A Placebo-Controlled Study Evaluating the Potential Effects of Trabectedin on the Heart in Patients with Advanced Cancer — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=789&filename=CR014917_CSR.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted in 7 countries: Belgium (3 sites), France (2 sites), India (2 sites), Republic of Korea (4 sites), Russia (4 sites), Spain (1 site), and the United States (4 sites). Total 75 participants were enrolled in this study.
Pre-assignment Details: All enrolled participants (ie, 75 participants) received study medication. 26 participants completed the study.
Groups:
- Trabectedin: 1.3 mg/m2 of trabectedin was administered as a 3-hour intravenous infusion on Day 2
Period: Overall Study
Arm/Group | Trabectedin
Started | 75
Completed | 26
Not Completed | 49
Not completed — Physician Decision | 4
Not completed — Death | 4
Not completed — Adverse Event | 6
Not completed — Progressive disease | 31
Not completed — Withdrawal by Subject | 4

BASELINE CHARACTERISTICS:
Arm/Group | Trabectedin
Number analyzed (Participants) | 75
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.2 (11.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51
  Male | 24
Race/Ethnicity, Customized [Number; unit: participants]
  White | 51
  Asian | 23
  Other | 1
Region of Enrollment [Number; unit: participants]
  Belgium | 17
  France | 3
  India | 8
  Republic Of Korea | 15
  Russia | 17
  Spain | 4
  United States Of America | 11

OUTCOME MEASURES:

1. Primary Outcome: The Difference in the Change From Baseline (Predose on Day 1) in QTc Intervals Trabectedin Relative to Placebo at 24 Hour Post Dose by Fridericia Correction
Description: QTc interval was measured by electrocardiograms to evaluate the potential effect of trabectedin on QTc interval duration. The Fridericia correction was used as the standard clinical correction for calculating the heart rate-corrected QT interval.
Time Frame: Baseline (predose on Day 1) to 24 hour post dose (Day 1 or Day 2)
Population: All evaluable participants set: All participants who received placebo on Day 1 and trabectedin on Day 2 with atleast 1 paired predose and 1 paired postdose assessments. One participant who received study medication in reverse order (trabectedin and placebo were given on Days 1 and 2, respectively) was excluded from evaluations.
Measure: Mean (Standard Deviation); unit: milli seconds
Groups:
- Placebo: Placebo: Normal saline was administered as a 3-hour intravenous infusion on Day 1.
Arm/Group | Placebo | Trabectedin
Number analyzed (Participants) | 74 | 74
milli seconds | 3.6 (10.08) | -6.2 (10.65)

2. Secondary Outcome: Maximum Plasma Concentration of Trabectedin (Cmax)
Time Frame: Baseline (predose on Day 2) to 24 hour post dose (Day 2 or Day 3).
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: nanogram per milliliter
Arm/Group | Trabectedin
Number analyzed (Participants) | 74
nanogram per milliliter | 9.24 (3.75)

3. Secondary Outcome: Time Taken to Acheive Maximum Plasma Concentration (Tmax)
Time Frame: Baseline (predose on Day 2) to 24 hour post dose (Day 2 or Day 3).
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Trabectedin
Number analyzed (Participants) | 74
hours | 2.22 (0.65)

4. Secondary Outcome: Number of Participants With QTc Interval Increase From Baseline (Predose on Day 1) Greater Than 30 Milli Seconds
Description: The Fridericia (QTcF) and Bazett's (QTcB) correction were used as the standard clinical correction for calculating the heart rate-corrected QT interval.
Time Frame: Baseline (predose) to approximately 24 hour post dose
Population: as for outcome 1
Measure: Number; unit: participants
Groups:
- Placebo: Normal saline was administered as a 3-hour intravenous infusion on Day 1
Arm/Group | Placebo | Trabectedin
Number analyzed (Participants) | 74 | 74
participants
  QTcF greater than 30 milliseconds | 2 | 2
  QTcB greater than 30 milliseconds | 4 | 6

5. Secondary Outcome: Number of Participants With QTc Interval Increase From Baseline (Predose on Day 1) Greater Than 60 Milli Seconds
Description: as for outcome 4
Time Frame: Baseline (predose) to approximately 24 hour post dose
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Placebo | Trabectedin
Number analyzed (Participants) | 74 | 74
participants
  QTcF greater than 60 milliseconds | 0 | 0
  QTcB greater than 60 milliseconds | 0 | 0

6. Secondary Outcome: Number of Participants With QTc Interval Greater Than 450 Milli Seconds
Description: as for outcome 4
Time Frame: Baseline (predose) to approximately 24 hour post dose
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Placebo | Trabectedin
Number analyzed (Participants) | 74 | 74
participants
  QTcF greater than 450 milliseconds | 6 | 4
  QTcB greater than 450 milliseconds | 21 | 23

7. Secondary Outcome: Number of Participants With QTc Interval Greater Than 480 Milli Seconds
Description: The Fridericia (QTcF) and Bazett's (QTcB) correction were used as the standard clinical correction for calculating the heart rate-corrected QTc interval.
Time Frame: Baseline (predose) to approximately 24 hour post dose
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Placebo | Trabectedin
Number analyzed (Participants) | 74 | 74
participants
  QTcF greater than 480 milli seconds | 0 | 0
  QTcB greater than 480 milli seconds | 1 | 2

8. Secondary Outcome: Number of Participants With QTc Interval Greater Than 500 Milli Seconds
Description: as for outcome 7
Time Frame: Baseline (predose) to approximately 24 hour post dose
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Placebo | Trabectedin
Number analyzed (Participants) | 74 | 74
participants
  QTcF greater than 500 milli seconds | 0 | 0
  QTcB greater than 500 milli seconds | 0 | 0

9. Secondary Outcome: Number of Participants With PR Interval Greater Than 200 Milli Seconds
Description: PR interval is the portion of the electrocardiogram between the onset of the P wave (atrial depolarization) and the QRS complex (ventricular depolarization).
Time Frame: Baseline (predose) to approximately 24 hour post dose
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Placebo | Trabectedin
Number analyzed (Participants) | 74 | 74
participants | 3 | 2

10. Secondary Outcome: Number of Participants With QRS Interval Greater Than 120 Milli Seconds
Description: QRS interval is the interval from the beginning of the Q wave to the termination of the S wave, representing the time for ventricular depolarization.
Time Frame: Baseline (predose) to approximately 24 hour post dose
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Placebo | Trabectedin
Number analyzed (Participants) | 74 | 74
participants | 1 | 1

11. Secondary Outcome: Mean Heart Rate (Beats Per Minute) Over 24 Hours Postdose
Time Frame: Baseline (predose on Day 1) to 24 hour post dose
Population: All evaluable participants set: All participants who received placebo on Day 1 and trabectedin on Day 2 with atleast 1 paired predose and 1 paired postdose assessments. One participant who received study medication in reverse order was excluded from evaluations. 73 participants analyzed in trabectedin group to derive the mean.
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Placebo | Trabectedin
Number analyzed (Participants) | 74 | 73
beats per minute | 76.9 (10.51) | 82.6 (11.13)

12. Primary Outcome: The Difference in the Change From Baseline (Predose on Day 1) in QTc Intervals Trabectedin Relative to Placebo at 24 Hour Post Dose by Bazett's Correction
Description: QTc interval was measured by electrocardiograms to evaluate the potential effect of trabectedin on QTc interval duration. The Bazett's Correction was used as the standard clinical correction for calculating the heart rate-corrected QT interval.
Time Frame: Baseline (predose on Day 1) to 24 hour post dose (Day 1 or Day 2)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: milli seconds
Arm/Group | Placebo | Trabectedin
Number analyzed (Participants) | 74 | 74
milli seconds | 0.1 (10.15) | -1.5 (13.61)

ADVERSE EVENTS:
Time Frame: Until 30 days after the administration of the last dose of study medication
Description: Adverse events were reported for overall study.
Arm/Group | Trabectedin
Serious Adverse Events (participants affected / at risk) | 31/75
Other Adverse Events (participants affected / at risk) | 70/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Trabectedin (N=75)
Anaemia (Blood and lymphatic system disorders) | 2
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 5
Leukopenia (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 6
Thrombocytopenia (Blood and lymphatic system disorders) | 4
Abdominal pain (Gastrointestinal disorders) | 1
Haematochezia (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Subileus (Gastrointestinal disorders) | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 4
Asthenia (General disorders) | 4
Disease progression (General disorders) | 1
Mucosal inflammation (General disorders) | 1
Pyrexia (General disorders) | 4
Hepatic function abnormal (Hepatobiliary disorders) | 2
Hypertransaminasaemia (Hepatobiliary disorders) | 1
Cellulitis (Infections and infestations) | 1
Infection (Infections and infestations) | 1
Oral fungal infection (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Wound infection (Infections and infestations) | 1
Tibia fracture (Injury, poisoning and procedural complications) | 1
Anorexia (Metabolism and nutrition disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 3
Soft tissue haemorrhage (Musculoskeletal and connective tissue disorders) | 1
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Bone sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Oropharyngeal cancer stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Syncope (Nervous system disorders) | 1
Hydronephrosis (Renal and urinary disorders) | 1
Renal failure (Renal and urinary disorders) | 2
Renal impairment (Renal and urinary disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Capillary leak syndrome (Vascular disorders) | 1
Embolism (Vascular disorders) | 1
Iliac artery occlusion (Vascular disorders) | 1
Vena cava thrombosis (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Trabectedin (N=75)
Anaemia (Blood and lymphatic system disorders) | 22
Leukopenia (Blood and lymphatic system disorders) | 9
Neutropenia (Blood and lymphatic system disorders) | 31
Thrombocytopenia (Blood and lymphatic system disorders) | 13
Abdominal pain (Gastrointestinal disorders) | 5
Abdominal pain upper (Gastrointestinal disorders) | 4
Constipation (Gastrointestinal disorders) | 8
Diarrhoea (Gastrointestinal disorders) | 5
Nausea (Gastrointestinal disorders) | 38
Vomiting (Gastrointestinal disorders) | 30
Asthenia (General disorders) | 24
Fatigue (General disorders) | 17
Oedema peripheral (General disorders) | 4
Pain (General disorders) | 4
Pyrexia (General disorders) | 8
Hepatic function abnormal (Hepatobiliary disorders) | 33
Anorexia (Metabolism and nutrition disorders) | 16
Enzyme abnormality (Metabolism and nutrition disorders) | 8
Hypocalcaemia (Metabolism and nutrition disorders) | 6
Myalgia (Musculoskeletal and connective tissue disorders) | 4
Dizziness (Nervous system disorders) | 12
Cough (Respiratory, thoracic and mediastinal disorders) | 8
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days